CLINICAL TRIAL: NCT02132013
Title: SodiUm Burden Lowered by Lifestyle Intervention: Self-Management and E-health Technology
Acronym: SUBLIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Kidney Foundation (Other); Leiden University Medical Center (Other); St. Antonius Hospital (Other); Ziekenhuisgroep Twente (Other); TNO (Other)
Responsible Party: Principal Investigator, prof.dr. G.J. Navis, prof.dr. G.J. Navis, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL48079.042.14; METC 2014/075 (Other: Medical Ethics Committee, UMCG); 837001005 (Other Grant/Funding Number: ZonMW)
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Kidney Disease; Unspecified Complication of Kidney Transplant
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention SUBLIME (Experimental): Intervention group
  Interventions: Behavioral: Intervention SUBLIME
- Control (No Intervention): Regular care

INTERVENTIONS:
Behavioral: Intervention SUBLIME — Intervention: dietary sodium restriction supported by 2 group meetings, structured self-regulation computer program, e-coaching.
  Arms: Intervention SUBLIME

SUMMARY:
The purpose of this study is to evaluate the effects and efficacy of dietary sodium restriction by mean of a new healthcare approach in patients with chronic kidney disease. The test persons in the intervention group are actively supported to adhere to a restricted sodium diet with a structured self-regulation program to implement sodium recommendations that are in current guidelines.

DETAILED DESCRIPTION:
The intervention entails two group meetings with fellow-patients, motivational interviewing, e-coaching and ICT-based self-regulation as add-on to regular care. The intervention consists of a baseline measurement (T0), followed by a preparation phase of 2-3 weeks duration before the first group meeting. The first group meeting is followed by the action phase with a second group meeting in 9-11 weeks. During the action phase, test persons are stimulated to use the special self-regulation computer program, monitor their dietary sodium intake on this website and receive e-coaching from their personal coach. Test persons in the control group receive standard care. After 3 months in study (T1), all test persons visit the outpatient clinic for measurements and data collection. The half year long maintenance phase starts after this timepoint, test persons in the intervention group can continue the use of the special website and get feedback from their coach at 3, 4, 5, 6 months. After 9 months of total study duration (T2), data collection and measurements take place.

At each timepoint blood and 24-hourly urine is collected, test persons fill out questionnaires. The intervention group collects after 5 weeks in study an additional 24-hourly urine collection to assess dietary compliance and enable feedback.

Cost-efficacy and implementation analysis will be conducted after study closure.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older.
* Have chronic kidney disease (CKD stage 1-3, CKD 4 if eGFR is not lower than 25 mL/min/1.73m2, or be a renal transplant recipient.)
* Have a urinary sodium excretion during at least the last 2 subsequent visits of more than 130 mmol per day, or one last urinary sodium excretion of more than 150 mmol per day.
* Have a systolic blood pressure higher than 135 mmHg, diastolic blood pressure higher than 85 mmHg or a well-controlled blood pressure by treatment with antihypertensives including RAAS-blockade (ACE-inhibitor or ARB).
* Sufficient command of the Dutch language.
* Access and ability to use the internet.
* Written informed consent.

Exclusion Criteria:

* eGFR < 25 ml/min/1.73m2 or an anticipated need for predialysis work-up within the time frame of the study.
* Unstable disease: defined as rapid, persistent, progressive renal function loss (e.g. > 6 mL/min/1.73m2 per year), not from acute, intermittent origin.
* Blood pressure > 170 mmHg systolic or > 100 mmHg diastolic during medical treatment
* Blood pressure < 95 mmHg systolic not responding to withdrawal of antihypertensives.
* Cardiovascular event (myocardial infarction, cerebrovascular accident) < 6 months ago.
* Renal transplantation <1 year ago.
* Medical conditions that are likely to interfere with completion of the study (such as progressive malignancy or other debilitating illness) at the discretion of the nephrologist.
* Every patient who has participated in the ESMO study (regardless whether intervention or control) cannot participate in the current study.
* Current participation in any clinical trial that might interfere with SUBLIME trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
24-hourly urinary sodium excretion | up to 9 months

SECONDARY OUTCOMES:
Blood pressure | 0, 3, 9 months
Psychological well-being | 0, 3, 9 months
  Psychological well-being will be assessed with multiple choice questionnaires in all 150 participants.
Cost-effectiveness | After study closure
  Cost-effectiveness will be calculated from data derived from questionnaires on health care use (contacts with health care professionals, change in medication) in all participants.

OTHER OUTCOMES:
Tertiary: effect of sodium restriction on cardiorenal biomarkers | 0, 3 or 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerjan J Navis, MD PhD, Study Chair — University Medical Center Groningen; Paul JM Van der Boog, MD PhD, Principal Investigator — Leiden University Medical Center; Sandra Van Dijk, PhD, Principal Investigator — Leiden University Medical Center
Locations (4):
- Netherlands (4):
  - Ziekenhuisgroep Twente, Almelo, Overijssel
  - University Medical Center Groningen, Groningen, Provincie Groningen
  - Leiden University Medical Center, Leiden, South Holland
  - St. Antonius, Nieuwegein, Utrecht

REFERENCES:
- [Derived] McMahon EJ, Campbell KL, Bauer JD, Mudge DW, Kelly JT. Altered dietary salt intake for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jun 24;6(6):CD010070. doi: 10.1002/14651858.CD010070.pub3. PMID 34164803
- [Derived] Humalda JK, Klaassen G, de Vries H, Meuleman Y, Verschuur LC, Straathof EJM, Laverman GD, Bos WJW, van der Boog PJM, Vermeulen KM, Blanson Henkemans OA, Otten W, de Borst MH, van Dijk S, Navis GJ; SUBLIME Investigators. A Self-management Approach for Dietary Sodium Restriction in Patients With CKD: A Randomized Controlled Trial. Am J Kidney Dis. 2020 Jun;75(6):847-856. doi: 10.1053/j.ajkd.2019.10.012. Epub 2020 Jan 16. PMID 31955921